CLINICAL TRIAL: NCT01498419
Title: A Phase II Open-Label Partially Randomized Trial to Evaluate the Efficacy, Safety and Tolerability of the Combination of Moxifloxacin Plus PA-824 Plus Pyrazinamide After 8 Weeks of Treatment in Adult Patients With Newly Diagnosed Drug-Sensitive or Multi Drug-Resistant, Smear-Positive Pulmonary Tuberculosis
Brief Title: Evaluation of 8 Weeks of Treatment With the Combination of Moxifloxacin, PA-824 and Pyrazinamide in Patients With Drug Sensitive and Multi Drug-Resistant Pulmonary Tuberculosis (TB) (NC-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NC-002-(M-Pa-Z)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2017-01

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; Serial Sputum Colony Counts; Colony Forming Units; Time to Sputum Culture Positivity; PA824; pretomanid
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Moxifloxacin; pretomanid; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) (Experimental): Drug Sensitive Participants: One moxifloxacin (M) 400 mg tablet plus one Pretomanid (PA-824) 100 mg tablet plus three pyrazinamide 500 mg tablets taken once daily for 8 weeks
  Interventions: Drug: Moxifloxacin (M); Drug: Pretomid (Pa); Drug: Pyrazinamide (Z)
- Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) (Experimental): Drug Sensitive Participants: One moxifloxacin (M) 400 mg tablet plus one Pretomanid (PA-824) 200 mg tablet plus three pyrazinamide 500 mg tablets taken once daily for 8 weeks
  Interventions: Drug: Moxifloxacin (M); Drug: Pretomid (Pa); Drug: Pyrazinamide (Z)
- Drug Sensitive: Rifafour (Active Comparator): Drug Sensitive Participants: Rifafour was administered orally once daily for 8 weeks according to weight: 30 kg to 37 kg: two tablets; 38 kg to 54 kg: three tablets; 55 kg to 70 kg: four tablets; ≥71 kg: five tablets
  Interventions: Drug: Rifafour
- Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg) (Experimental): Multi Drug-Resistant Participants: One moxifloxacin (M) 400 mg tablet plus one Pretomanid (PA-824) 200 mg tablet plus three pyrazinamide 500 mg tablets taken once daily for 8 weeks
  Interventions: Drug: Moxifloxacin (M); Drug: Pretomid (Pa); Drug: Pyrazinamide (Z)

INTERVENTIONS:
Drug: Moxifloxacin (M)
  Arms: Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg); Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg); Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Drug: Pretomid (Pa)
  Other Names: PA-824
  Arms: Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg); Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg); Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Drug: Pyrazinamide (Z)
  Arms: Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg); Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg); Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Drug: Rifafour — Rifafour e-275 once daily for 8 weeks. Daily dose dependent on weight as follows: 30-37kg: 2 tablets, 38-54 kg: 3 tablets, 55-70 kg: 4 tablets: 71 kg and over: 5 tablets
  Arms: Drug Sensitive: Rifafour

SUMMARY:
The purpose of this study is to assess the mycobactericidal activity of the moxifloxacin plus PA-824 plus pyrazinamide regimen after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all trial-related procedures including HIV testing (if an HIV test was performed within 1 month prior to trial start, it should not be repeated as long as documentation can be provided [ELISA and/or Western Blot]).
* Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
* Sputum smear-positive pulmonary TB (at trial appointed laboratory). For Drug Sensitive TB treatment arms, subjects should be newly diagnosed and previously untreated. Exception: Participants can be included in the trial if they were diagnosed and treated for TB greater than 5 years prior to screening and can provide documentation of cure for that episode. Additionally, participants who have previously received H prophylactically can be included as long as that treatment is/was discontinued at least 7 days prior to randomization into this trial. Drug sensitive status to be confirmed with fluoroquinolone, rifampicin and isoniazid susceptibility testing at screening using Hain Plus rapid sputum test.

For the MDR-TB treatment arm only: Subjects with smear-positive MDR infection, defined as confirmed resistance to at least both R and H confirmed at screening for entry into this trial. Resistance to R and H will be determined using the rapid screen test (Hain Plus). If the first spot sputum shows an indeterminate result, the test must be repeated on freshly collected spot sputum or overnight sputum and that result may be used.

Subjects with newly diagnosed MDR-TB are defined as a) subjects with MDR-TB who have never been treated for TB before, or b) subjects with MDR-TB who have previously been treated with only one course of first-line TB drugs (H, R, E, Z and/or S) and that treatment is/was discontinued at least 7 days prior to randomization into this trial. Additionally, MDR-TB participants who have previously received H prophylactically can be included as long as that treatment is/was discontinued at least 7 days prior to randomization into this trial.

* A chest X-ray picture which in the opinion of the Investigator is compatible with TB.
* Sputum positive (at site laboratory) on direct microscopy for acid-fast bacilli (at least 1+ on the IUATLD/WHO scale).
* Ability to produce an adequate volume of sputum as estimated from a spot assessment (estimated 10 ml or more overnight production).
* Females may participate if they are: 1) of non-childbearing potential (have had a bilateral oophorectomy, tubal ligation and/or hysterectomy or have been postmenopausal for at least 12 consecutive months), 2) if they are using effective birth control methods and are willing to continue practicing birth control methods throughout treatment or 3) be non-heterosexually active, practice sexual abstinence or have a vasectomized partner (confirmed sterile). Therefore to be eligible for this study women of childbearing potential should either: 1) use a double barrier method to prevent pregnancy (i.e. use a condom with either diaphragm or cervical cap) or 2) use hormonal based contraceptives in combination with a barrier contraceptive, or 3) use an intrauterine device in combination with a barrier contraceptive. They must also be willing to continue these contraceptive measures until one week after the last dose of study medication or one week after discontinuation from study medication in case of premature discontinuation. (Note: Hormone-based contraception alone may not be reliable when taking IMP; therefore, hormone-based contraceptives alone cannot be used by female participants to prevent pregnancy).
* Male participants who are having heterosexual intercourse with females of child-bearing potential are required to use one of the following birth control methods during their participation in the trial and for 12 weeks after their last dose of study medication to prevent pregnancy:
* a double barrier method which can include a male condom, diaphragm, cervical cap, or female condom; or
* a barrier method combined with hormone-based contraceptives or an intra-uterine device for the female partner.

The use of the above mentioned birth control method does not apply if the male participant has been vasectomised or has had a bilateral orchidectomy minimally three months prior to screening, or is not heterosexually active, or practices sexual abstinence or if the female sexual partner has had a bilateral oophorectomy, tubal ligation and/or hysterectomy or has been postmenopausal for at least 12 consecutive months.

Exclusion Criteria:

* Evidence of clinically significant (as judged by the investigator), metabolic, gastrointestinal, cardiovascular, musculoskeletal, ophthalmological, pulmonary, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied) including myasthenia gravis and malaria.
* End stage liver failure (class Child Pugh C).
* Poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
* Clinically significant evidence of extrathoracic TB (e.g. miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator.
* History of allergy or hypersensitivity to any of the study IMP or related substances, including a known allergy to any fluoroquinolone antibiotic, history of tendinopathy associated with quinolones or suspected hypersensitivity to any rifamycin antibiotics.
* Resistance to fluoroquinolones (Hain plus rapid test) and/or pyrazinamide. Participants may be included in the study prior to receipt of the susceptibility test results for fluoroquinolones or pyrazinamide, however once these are received after a participant has entered into the study and if the results show the participant is resistant to fluoroquinolones and/or pyrazinamide, such a participant should be removed from the trial. DS participants will not be replaced, but MDR-TB participants taking part in the EBA Sub-Study could be replaced after consultation and written approval with the sponsor.
* Known (positive urine drug screen) or suspected, current or history of within the past 2 years, alcohol or drug abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the participant.
* For HIV infected participants:
* having a CD4+ count <200 cells/µL;
* or having received intravenous antifungal medication within the last 90 days;
* or with an AIDS-defining opportunistic infection or malignancies (except pulmonary TB).
* Having participated in other clinical study/ies with investigational agent/s within 8 weeks prior to trial start.
* Significant cardiac arrhythmia requiring medication.
* Participants with the following at screening (per measurements and reading done by Central ECG):
* Marked prolongation of QT/QTc interval, e.g., confirmed demonstration of QTcF (Fridericia correction) or QTcB (Bazett correction) interval >450 ms at screening;
* History of additional risk factors for Torsade de Pointes, e.g., heart failure, hypokalemia, family history of Long QT Syndrome;
* Use of concomitant medications that are known to prolong the QT/QTc interval (see exclusion criterion 21 as well as list of disallowed medication in the study protocol);
* Any clinically significant, in the opinion of the Investigator, ECG abnormality.
* Females who are pregnant, breast-feeding, or planning to conceive a child within one week of cessation of treatment.
* Males planning to conceive a child within twelve weeks of cessation of treatment.
* History and/or presence (or evidence) of neuropathy or epilepsy.
* Diabetes Mellitus requiring insulin.
* History of lens opacity or evidence of lens opacity on slit lamp ophthalmologic examination.
* Previously received treatment with PA-824 as part of a clinical trial.
* For the DS-TB treatment arms: treatment with any drug active against MTB within the 3 months prior to Visit 1 (e.g. isoniazid, ethambutol, amikacin, clofazimine, cycloserine, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, fluoroquinolones, thioamides, metronidazole). Exceptions noted in Inclusion Criteria.
* For the MDR-TB Subjects: previously treated for MDR-TB. Defined as having received multiple courses of first-line therapy or any second-line TB drug, including any of the following anti-mycobacterials: any aminoglycoside except streptomycin, any fluoroquinolone, the thioamides, prothionamide or ethionamide and cycloserine.
* Any diseases or conditions in which the use of the standard TB drugs or any of their components is contra-indicated, including but not limited to allergy to any TB drug, their component or to the IMP.
* Any disease or conditions in which any of the medicinal products listed in the section of the protocol pertaining to prohibited medications is used.
* Use of any drug within 30 days prior to dosing known to prolong QTc interval (including amiodarone, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, sotalol, sparfloxacin, thioridazine). Exceptions may be made for participants that have received 3 days or less of one of these drugs or substances, if there has been a wash-out period before administration of IMP equivalent to at least 5 half-lives of that drug or substance.
* Use of any therapeutic agents known to alter any major organ function (e.g., barbiturates, opiates, phenothiazines, cimetidine) within 30 days prior to dosing. The Investigator may choose at his/her discretion to make an exception for opiates or painkillers if they were part of prescribed medication for cough or underlying disease.
* Use of systemic glucocorticoids within one year prior to dosing.
* Participants with the following toxicities at screening as defined by the enhanced Division of Microbiology and Infectious Disease (DMID) adult toxicity table (November 2007):
* creatinine grade 2 or greater (>1.5 times upper limit of normal [ULN]);
* creatinine clearance (CrCl) level less than 30 mls/min. according to the Cockcroft-Gault Formula;
* hemoglobin grade 4 (<6.5 g/dL);
* platelets grade 2 or greater (under 50x109 cells/L);
* serum potassium less than the lower limit of normal for the laboratory;
* aspartate aminotransferase (AST) grade 3 or greater (≥3.0 x ULN) to be excluded;
* alanine aminotransferase (ALT) grade 3 or greater (≥3.0 x ULN) to be excluded;
* alkaline phosphatase (ALP) grade 4 (>8.0 x ULN) to be excluded, grade 3 (≥3.0 - 8.0 x ULN) must be discussed with the sponsor Medical Monitor;
* total bilirubin grade 3 or greater (>2.0 x ULN, or >1.50 x ULN when accompanied by any increase in other liver function test) to be excluded, grade 2 (>1.50 x ULN, or >1.25 x ULN when accompanied by any increase in other liver function test) must be discussed with the sponsor Medical Monitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Dawson, MD, Principal Investigator — University of Cape Town
Locations (8):
- South Africa (6):
  - Task Applied Science, Karl Bremer Hospital, Cape Town
  - University of Cape Town Lung Institute (Pty) Ltd, Cape Town
  - KwaZulu-Natal Research Institute for Tuberculosis and HIV (K-RITH), Durban
  - CHRU Themba Lethu Clinic, Johannesburg
  - Klerksdorp Tshepong Hospital, Klerksdorp
  - The Aurum Institute: Tembisa Hospital, Tembisa
- Tanzania (2):
  - Ifakara Health Institute, Bagamoyo
  - Mbeya Medical Research Programme, Mbeya

REFERENCES:
- [Result] Dawson R, Diacon AH, Everitt D, van Niekerk C, Donald PR, Burger DA, Schall R, Spigelman M, Conradie A, Eisenach K, Venter A, Ive P, Page-Shipp L, Variava E, Reither K, Ntinginya NE, Pym A, von Groote-Bidlingmaier F, Mendel CM. Efficiency and safety of the combination of moxifloxacin, pretomanid (PA-824), and pyrazinamide during the first 8 weeks of antituberculosis treatment: a phase 2b, open-label, partly randomised trial in patients with drug-susceptible or drug-resistant pulmonary tuberculosis. Lancet. 2015 May 2;385(9979):1738-1747. doi: 10.1016/S0140-6736(14)62002-X. Epub 2015 Mar 18. PMID 25795076

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg): Drug Sensitive Participants received moxifloxacin (M) (one 400 mg tablet), pretomanid (Pa-824; Pa) (one 100 mg tablet), and pyrazinamide (Z) (three 500 mg tablets) once daily for 8 weeks
- Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg): Drug Sensitive Participants received moxifloxacin (M) (one 400 mg tablet), pretomanid (Pa-824; Pa) (one 200 mg tablet), and pyrazinamide (Z) (three 500 mg tablets) once daily for 8 weeks
- Drug Sensitive: Rifafour: Drug Sensitive Participants received Rifafour e-275 once daily for 8 weeks. Daily dose dependent on weight as follows: 30-37kg: two tablets, 38-54kg: three tablets, 55-70kg: four tablets: 71kg and over: five tablets
- Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg): Multi Drug-Resistant Participants received moxifloxacin (M) (one 400 mg tablet), pretomanid (Pa-824; Pa) (one 200 mg tablet), and pyrazinamide (Z) (three 500 mg tablets) once daily for 8 weeks
Period: Overall Study
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Started | 60 | 62 | 59 | 26
Completed | 42 | 39 | 41 | 7
Not Completed | 18 | 23 | 18 | 19

BASELINE CHARACTERISTICS:
Population: The ages of four participants in the Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) group and one participant in the Drug Sensitive: Rifafour group were missing and so were not included in the demographics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg) | Total
Number analyzed (Participants) | 60 | 62 | 59 | 26 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Analysis Population
  years | 29.5 (10.63) | 30.9 (8.96) | 30.4 (9.75) | 32.4 (9.75) | 30.6 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Analysis Population
  Participants
    Female | 22 | 22 | 18 | 10 | 72
    Male | 38 | 40 | 41 | 16 | 135
Race/Ethnicity, Customized [Number; unit: participants] — Safety Analysis Population
  participants
    Black | 43 | 46 | 43 | 15 | 147
    Mixed Ethnic | 17 | 16 | 16 | 11 | 60
Weight [Mean (Standard Deviation); unit: kilograms] — Safety Analysis Population
  kilograms | 54.7 (8.72) | 57.6 (10.09) | 54.7 (7.95) | 57.9 (10.61) | 56 (9.25)
HIV Status [Number; unit: participants] — Safety Analysis Population
  participants
    Positive | 12 | 8 | 13 | 7 | 40
    Negative | 48 | 53 | 45 | 18 | 164
    Indeterminate | 0 | 0 | 1 | 0 | 1
    Missing | 0 | 1 | 0 | 1 | 2
Pyrazinamide susceptibility [Number; unit: participants] — Safety Analysis Population
  participants
    Resistant | 0 | 2 | 1 | 17 | 20
    Sensitive | 60 | 59 | 58 | 9 | 186
    Missing | 0 | 1 | 0 | 0 | 1
Moxifloxacin susceptibility [Number; unit: participants] — Safety Analysis Population
  participants
    Resistant | 0 | 2 | 1 | 1 | 4
    Sensitive | 56 | 58 | 57 | 25 | 196
    No Result | 3 | 2 | 1 | 0 | 6
    Unclear | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Change in Colony Forming Units (CFUs) Using Non-linear Mixed Effects Modeling of the Serial Sputum Colony Counts (SSCC) Over 8 Weeks of Treatment.
Description: The primary efficacy endpoint was bactericidal activity characterized by the daily rate of change in mean log10CFU counts during 8 weeks of treatment (bactericidal activity assessed by CFU on solid media for days 0-56).
Time Frame: 8 weeks
Population: The efficacy analysis population contained patients included in the safety analysis population for whom efficacy data were available and who had no major protocol violations that could affect the integrity of the efficacy data. The number of participants analyzed for this outcome was 173.
Measure: Mean (95% Confidence Interval); unit: log10CFU/ml/day
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Number analyzed (Participants) | 56 | 54 | 54 | 9
log10CFU/ml/day | 0.133 [0.109 to 0.155] | 0.155 [0.133 to 0.178] | 0.112 [0.093 to 0.131] | 0.117 [0.070 to 0.174]

2. Secondary Outcome: Time to Sputum Conversion Using Data From Weekly Cultures Through 8 Weeks on Liquid Media
Description: liquid culture = Mycobacteria growth indicator tube (MGIT) Sputum culture conversion is defined as a change from a positive growth of M. tuberculosis in a sputum sample to negative M. tuberculosis growth sputum sample in patients with pulmonary TB
Time Frame: 8 weeks
Population: The efficacy analysis population contained participants included in the safety analysis population for whom efficacy data were available and who had no major protocol violations that could affect the integrity of the efficacy data. The number of participants included for this outcome was 206.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Number analyzed (Participants) | 60 | 61 | 59 | 26
days | 42.0 [35.0 to NA] — There were not enough conversion events to determine the 75th percentile | 49.0 [41.0 to 56.0] | 56.0 [43.0 to NA] — There were not enough conversion events to determine the 75th percentile | 56.0 [45.0 to NA] — There were not enough conversion events to determine the 75th percentile

3. Secondary Outcome: Percentage of Patients With Sputum Culture Conversion at 8 Weeks on Solid Media
Description: Sputum culture conversion is defined as a change from a positive growth of M. tuberculosis in a sputum sample to negative M. tuberculosis growth sputum sample in patients with pulmonary TB. (Day 57)
Time Frame: Day 57 after eight weeks of daily treatment
Population: The efficacy analysis population contained participants included in the safety analysis population for whom efficacy data were available and who had no major protocol violations that could affect the integrity of the efficacy data. Participants included in this outcome had a valid, non-contaminated culture from the sample acquired on Day 57.
Measure: Number; unit: percentage of participants
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Number analyzed (Participants) | 35 | 35 | 32 | 8
percentage of participants | 82.9 | 94.3 | 87.5 | 62.5

4. Secondary Outcome: The Rate of Change in Time to Sputum Culture Positivity (TTP) Through 8 Weeks in the MGIT System in Sputum Over 8 Weeks in Participants as Derived From a Non-linear Regression Model.
Description: Measurement of TTP in liquid culture media Mycobacteria growth indicator tube (MGIT) using standard procedures
Time Frame: 8 weeks
Population: The efficacy analysis population contained patients included in the safety analysis population for whom efficacy data were available and who had no major protocol violations that could affect the integrity of the efficacy data. The number of participants analyzed for this outcome was 179.
Measure: Mean (95% Confidence Interval); unit: log10hours/day
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Number analyzed (Participants) | 55 | 57 | 58 | 9
log10hours/day | 0.020 [0.015 to 0.025] | 0.020 [0.016 to 0.024] | 0.017 [0.013 to 0.021] | 0.015 [-0.001 to 0.031]

5. Secondary Outcome: Percentage of Participants Who Discontinue Due to an Adverse Event in Each Experimental Arm.
Time Frame: 8 weeks
Population: The Safety population was analyzed for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Number analyzed (Participants) | 60 | 62 | 59 | 26
percentage of participants | 13 | 19 | 12 | 12

6. Secondary Outcome: Time to Sputum Conversion Using Data From Weekly Cultures Through 8 Weeks on Solid Media
Description: Sputum culture conversion is defined as a change from a positive growth of M. tuberculosis in a sputum sample to negative M. tuberculosis growth sputum sample in patients with pulmonary TB
Time Frame: 8 weeks
Population: The efficacy analysis population contained patients included in the safety analysis population for whom efficacy data were available and who had no major protocol violations that could affect the integrity of the efficacy data. The number of participants analyzed for this outcome was 206.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Number analyzed (Participants) | 60 | 61 | 59 | 26
days | 28.0 [14.0 to 35.0] | 28.0 [21.0 to 35.0] | 35.0 [21.0 to 49.0] | 35.0 [24.5 to 56.0]

7. Secondary Outcome: Percentage of Patients With Sputum Culture Conversion at 8 Weeks on Liquid Media
Description: Sputum culture conversion is defined as a change from a positive growth of M. tuberculosis in a sputum sample to negative M. tuberculosis growth sputum sample in patients with pulmonary TB. This was measured at visit 24(Day 57).
Time Frame: Day 57 after eight weeks of daily treatment
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Number analyzed (Participants) | 35 | 35 | 37 | 8
percentage of patients | 65.7 | 71.4 | 37.8 | 50.0

ADVERSE EVENTS:
Arm/Group | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) | Drug Sensitive: Rifafour | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg)
Serious Adverse Events (participants affected / at risk) | 1/60 | 7/62 | 1/59 | 0/26
Other Adverse Events (participants affected / at risk) | 52/60 | 57/62 | 50/59 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) (N=60) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) (N=62) | Drug Sensitive: Rifafour (N=59) | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg) (N=26)
Death - Cause Unknown (General disorders) | 1 | 0 | 0 | 0
Drug-Induced Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cardiac Arrhythmia (2nd degree AV block) (Cardiac disorders) | 0 | 1 | 0 | 0
Hyperuriceamia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Closed Tibia Plateau Fracture-Left Knee Joint (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Elevated Liver Enzymes (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Epileptic Seizures (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Liver Drug-Induced Toxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug Sensitive: M (400 mg) Pa (100 mg) Z (1500 mg) (N=60) | Drug Sensitive: M (400 mg) Pa (200 mg) Z (1500 mg) (N=62) | Drug Sensitive: Rifafour (N=59) | Multi Drug-Resistant: M (400 mg) Pa (200 mg) Z (1500 mg) (N=26)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 17 | 17 | 17 | 8
HYPONATRAEMIA (Metabolism and nutrition disorders) | 8 | 5 | 8 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4 | 2 | 3 | 3
ENZYME ABNORMALITY (Metabolism and nutrition disorders) | 2 | 4 | 4 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 4 | 2 | 5 | 0
NAUSEA (Gastrointestinal disorders) | 14 | 8 | 7 | 8
VOMITING (Gastrointestinal disorders) | 7 | 7 | 7 | 4
DIARRHOEA (Gastrointestinal disorders) | 4 | 3 | 3 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 | 2 | 3 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 20 | 18 | 11 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 5 | 2 | 5 | 1
LIVER DISORDER (Hepatobiliary disorders) | 16 | 14 | 9 | 3
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 5 | 4 | 3 | 0
DIZZINESS (Nervous system disorders) | 6 | 8 | 2 | 1
HEADACHE (Nervous system disorders) | 6 | 6 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator or any Sub-Investigator shall submit any oral or written publication or abstract concerning this study to the Sponsor not less than thirty (30) days prior to submission to any journal, other publication or meeting, for review and removal of confidential information.